CLINICAL TRIAL: NCT05095519
Title: Hepatocellular Carcinoma Imaging Using PSMA PET/CT - a Prospective Pilot Trial
Brief Title: Hepatocellular Carcinoma Imaging Using PSMA PET/CT
Acronym: HepaSMART
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HREC/62461/PMCC
Record Dates: First submitted 2021-09-21; First posted 2021-10-27 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; PSMA; 18F-DCFPyL
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 18F-DCFPyL (Experimental): Patients will undergo PET/CT imaging following intravenous administration of 18F-DCFPyL
  Interventions: Drug: 18F-DCFPyL

INTERVENTIONS:
Drug: 18F-DCFPyL — 18F-DCFPyL will be administered with a single dose of 3.5 MBq per kg (2-4 MBq per kg), maximum 400 MBq), administered as a slow (over 30 seconds) intravenous injection

SUMMARY:
The purpose of the research is to evaluate the use of a PSMA PET/CT (Prostate Specific Membrane Antigen Positron Emission Tomography/Computerized Tomography) scan in the diagnosis of HCC (hepatocellular carcinoma) and comparing it to standard scanning techniques with CT (Computed Tomography) or MRI (Magnetic Resonance Imaging).

DETAILED DESCRIPTION:
A total of 30 patients will be recruited in this prospective pilot study who have HCC on imaging criteria (LI-RADS 5) for surgical resection, or patients with indeterminate liver lesions (LI-RADS 3 or 4) planned for liver biopsy. 18F-DCFPYL PSMA PET/CT will be performed prior to the planned surgery or liver biopsy

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or older at screening
* Has provided written informed consent for participation in the study
* Must have risk factors for HCC e.g. cirrhosis, chronic hepatitis B infection with or without cirrhosis
* Patients with liver lesions ≥1 cm suspicious for HCC but with indeterminate features on CT and MRI meeting LI-RADS 3 or 4 criteria planned for biopsy, OR patients with liver lesions diagnostic of HCC based on CT or MRI meeting LI-RADS 5 criteria planned for surgical resection
* Patients must be willing and able to comply with the protocol and procedures for the duration of the study
* Patients must be available for follow-up

Exclusion Criteria:

* Abdominal surgery or radiotherapy to the abdomen within <4 weeks of registration. Patients must have recovered from any effects of any major surgery
* Uncontrolled intercurrent illness that is likely to impede participation and or compliance
* Any history of prostate cancer or elevated PSA level for male patients
* Other malignancies unless curatively treated with no evidence of disease within previous 3-years other than adequately treated non-melanoma skin cancer or melanoma in situ
* Participation in another clinical study with an investigational product or another systemic cancer therapy administered in the last 4 weeks
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with requirements of the study
* Women who are pregnant or lactating
* Cirrhosis due to congenital hepatic fibrosis, vascular disorders (e.g. Budd-Chiari syndrome) or cardiac cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-08 (Actual); Primary Completion 2026-03-08 (Estimated); Study Completion 2026-09-08 (Estimated)

PRIMARY OUTCOMES:
True Positive Rate per patient | 6 months
  The probability that HCC is present when the PSMA-PET/CT test result is positive on a per patient basis.
True Negative Rate per patient | 6 months
  The probability that HCC is absent when the PSMA-PET/CT test result is negative on a per patient basis.
True Positive Rate per lesion | 6 months
  The probability that HCC is present when the PSMA-PET/CT test result is positive on a per lesion basis.
True Negative Rate per lesion. | 6 months
  The probability that HCC is absent when the PSMA-PET/CT test result is negative on a per lesion basis.

SECONDARY OUTCOMES:
PSMA uptake | 6 months
  Qualitative uptake of PSMA measured on a per lesion basis.
Maximum standard uptake value | 6 months
  Maximum standard uptake value of lesions on PSMA PET/CT.
CT LIRADS (Liver Imaging Reporting and Data System) Score | 6 months
  LI RADS Score for CT lesions.
PSMA expression. | 6 months
  Expression of PSMA per lesion.
GLUT-1 expression | 6 months
  Expression of GLUT 1 per lesion.

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - St Vincent's Hospital, Fitzroy, Victoria
  - Austin Health, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - The Royal Melbourne Hospital, Melbourne, Victoria